CLINICAL TRIAL: NCT02600117
Title: The Use of Tenofovir Disoproxil Fumarate (TDF) in the Management of Patients With Inactive Chronic Hepatitis B (CHB) Infection
Brief Title: Use of TDF in Patients With Inactive Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Florence Wong, MD, Hepatologist, Professor-Division of Gastroenterology,Department of Medicine, University of Toronto, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-8950; IN-CA-174-1708 (Other: Gilead Sciences, Inc.)
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir disoproxil fumarate (Other): 300 mg, orally, once a day for 3 years or when sAg+ve seroconverts to sAb+ve whichever comes earlier
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — 300 mg, oral, once a day
  Other Names: Viread

SUMMARY:
Recent evidence suggests that patients with inactive chronic hepatitis B (CHB) may develop the same types of liver complications that patients in the active state of hepatitis B virus (HBV) infection experience. Treatment guidelines for patients in the active state of HBV infection indicate that HBsAg clearance is associated with definitive remission of the activity of chronic HBV & improved long-term outcome. Clinical data showed that HBsAg clearance is achievable, in a small population of patients on continuous treatment with potent oral antivirals (OAVs), such as tenofovir disoproxil fumarate (TDF). It is possible the same OAVs can have the same effect in patients with inactive CHB, but in a shorter treatment duration. The purpose of this study is to find out if TDF is effective in controlling HBV DNA & promoting seroconversion from HBsAg-positive to HBsAb-positive in patients with inactive CHB.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a major worldwide health problem. The course of the majority of patients with inactive chronic hepatitis B is usually benign; therefore, the current treatment guidelines recommend not treating these patients. However, recent evidence suggests that the prognosis of these inactive carrier is not exactly benign. For instance, patients may develop liver cancer despite their inactive carrier state. Also, approximately 20-30% of patients with inactive chronic hepatitis B may undergo spontaneous reactivation of hepatitis over time. Multiple episodes of reactivation or sustained reactivation can cause progressive liver damage and even liver decompensation. However, until there are data to support that treatment with oral antivirals can alter the outcome of these patients, they will remain untreated. Potent oral antivirals have been shown to suppress HBV DNA and normalize liver enzymes in patients with active chronic hepatitis B infection. With continued long-term treatment, some of these patients have gone on to clear hepatitis B surface antigen and develop hepatitis B surface antibody. Therefore, it is possible that the same oral antivirals can have the same effect in patients with inactive chronic hepatitis B, but in a shorter duration of treatment. This study will explore the possible use of tenofovir disoproxil fumarate in controlling HBV DNA and promoting hepatitis B surface antigen seroconversion in patients with inactive chronic hepatitis B.

After completion of all initial investigations, patients will be started on TDF 300mg daily. Patients will be reviewed at 6 monthly intervals as per standard of care. At each clinic visit, patients will have blood tests including complete blood count, renal function, electrolytes, liver enzyme and liver function tests, as well as HBV serology including quantitative HBsAg and HBV DNA. Patients will also receive an abdominal ultrasound, fibroscan and fibrotest on an annual basis. Treatment will be stopped when sAg+ve seroconverts to sAb+ve or at the end of 3 years whichever comes earlier.

ELIGIBILITY:
Inclusion Criteria:

* All patients with inactive chronic hepatitis B, defined as someone who has HBV DNA ≤ log4, eAg-ve, eAb+, HBsAg+ve and normal ALT persistently for >6 months

Exclusion Criteria:

* Patients older than 75 years of age
* Presence of hepatoma at entry
* Presence of decompensated cirrhosis defined by a history of variceal bleed, ascites, or hepatic encephalopathy
* Presence of abnormal renal function defined as serum creatinine of>110µmol/L
* co-infection with HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Seroconversion from hepatitis B surface antigen positive to hepatitis B surface antibody positive | Three years
  Positive hepatitis B surface antibody result will indicate recovery from chronic hepatitis B virus infection.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Wong, MD, Principal Investigator — University Health Network -Toronto General Hospital
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada